CLINICAL TRIAL: NCT00899743
Title: Determining the Clinicopathological Significance of CaMKIIgamma Activation in AML
Brief Title: S9333A Study of Blood and Bone Marrow Samples From Patients With Previously Untreated Primary Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: S9333A; U10CA032102 (NIH); SWOG-9333A (Other: SWOG)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Leukemia
Keywords: adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); adult acute megakaryoblastic leukemia (M7); adult acute minimally differentiated myeloid leukemia (M0); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute myelomonocytic leukemia (M4); adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; untreated adult acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Congenital Abnormalities | interventions — Electrophoresis, Polyacrylamide Gel; Blotting, Western; Immunologic Techniques

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: polyacrylamide gel electrophoresis — polyacrylamide gel electrophoresis
Genetic: western blotting — western blotting
Other: immunologic technique — immunologic technique
Other: laboratory biomarker analysis — laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood and bone marrow from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is looking at blood and bone marrow samples from patients with previously untreated primary acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether calmodulin-dependent protein kinase II-γ (CaMKIIγ) activation (autophosphorylation) is associated with specific clinicopathological variables and outcomes in blood and bone marrow samples from patients with previously untreated primary acute myeloid leukemia.

OUTLINE: Blood and bone marrow samples are analyzed by western blot using SDS-PAGE and immunoblotting using anti-calmodulin-dependent protein kinase II-γ (CaMKIIγ) and anti-phosphospecific (Thr286, 287) CaMKIIγ antibodies with signals detected via chemiluminescence. CaMKIIγ activation levels are linked to clinical variables within the SWOG database.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Cryopreserved specimens of marrow or peripheral blood from patients enrolled in clinical trial SWOG-9333 and meeting the following criteria:

  * Diagnosis of primary acute myeloid leukemia

    * No M3 disease
    * Previously untreated disease
  * Randomized to remission induction chemotherapy with mitoxantrone hydrochloride and etoposide (Arm II)

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: specimens from S9333
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2008-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Association of specific clinicopathological variables and outcomes with calmodulin-dependent protein kinase II-γ (CaMKIIγ) activation (autophosphorylation) | upon receipt of specimens

CONTACTS AND LOCATIONS:
Overall Officials: Steven J. Collins, MD, Principal Investigator — Fred Hutchinson Cancer Center

REFERENCES:
- [Derived] Medeiros BC, Othus M, Fang M, Appelbaum FR, Erba HP. Cytogenetic heterogeneity negatively impacts outcomes in patients with acute myeloid leukemia. Haematologica. 2015 Mar;100(3):331-5. doi: 10.3324/haematol.2014.117267. Epub 2014 Dec 19. PMID 25527568
- [Derived] Medeiros BC, Othus M, Estey EH, Fang M, Appelbaum FR. Unsuccessful diagnostic cytogenetic analysis is a poor prognostic feature in acute myeloid leukaemia. Br J Haematol. 2014 Jan;164(2):245-50. doi: 10.1111/bjh.12625. Epub 2013 Oct 28. PMID 24383844